CLINICAL TRIAL: NCT05018871
Title: Safety of Cultured Autologous Adult Adipose Derived Mesenchymal Stem Cell Intravenous Infusion for the Treatment of Cerebral Palsy
Brief Title: Safety of Cultured Autologous Adult Adipose Derived Mesenchymal Stem Cell Intravenous Infusion for CP
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Covid-19
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-8-GR-8-04
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; CP; stem cell treatment
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Single intravenous infusion of 100 million cells
  Interventions: Biological: autologous adipose derived mesenchymal stem cells

INTERVENTIONS:
Biological: autologous adipose derived mesenchymal stem cells — cultured autologous adult adipose derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous infusion of cultured autologous adult adipose derived mesenchymal stem cells for the treatment of Cerebral Palsy

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of Cerebral Palsy (CP). This patient funded trial aims to study the safety and efficacy of intravenous infusion of cultured autologous adult adipose derived mesenchymal stem cells (AD-MSCs) for the treatment of CP. Patients with CP will receive a single intravenous infusion of AD-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cerebral Palsy

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety
* Previous organ transplant
* Seizure disorder
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: Gross Motor Function Measure (GMFM) | Four year follow-up
  It will be completed for each follow up point

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Mitera Hospital Athens Greece, Marousi, Greece

REFERENCES:
- [Background] Alotaibi M, Long T, Kennedy E, Bavishi S. The efficacy of GMFM-88 and GMFM-66 to detect changes in gross motor function in children with cerebral palsy (CP): a literature review. Disabil Rehabil. 2014;36(8):617-27. doi: 10.3109/09638288.2013.805820. Epub 2013 Jun 26. PMID 23802141
- [Background] Ko J, Kim M. Reliability and responsiveness of the gross motor function measure-88 in children with cerebral palsy. Phys Ther. 2013 Mar;93(3):393-400. doi: 10.2522/ptj.20110374. Epub 2012 Nov 8. PMID 23139425
- [Background] Huang L, Zhang C, Gu J, Wu W, Shen Z, Zhou X, Lu H. A Randomized, Placebo-Controlled Trial of Human Umbilical Cord Blood Mesenchymal Stem Cell Infusion for Children With Cerebral Palsy. Cell Transplant. 2018 Feb;27(2):325-334. doi: 10.1177/0963689717729379. PMID 29637820
- [Background] Min K, Song J, Kang JY, Ko J, Ryu JS, Kang MS, Jang SJ, Kim SH, Oh D, Kim MK, Kim SS, Kim M. Umbilical cord blood therapy potentiated with erythropoietin for children with cerebral palsy: a double-blind, randomized, placebo-controlled trial. Stem Cells. 2013 Mar;31(3):581-91. doi: 10.1002/stem.1304. PMID 23281216
- [Background] Liu X, Fu X, Dai G, Wang X, Zhang Z, Cheng H, Zheng P, An Y. Comparative analysis of curative effect of bone marrow mesenchymal stem cell and bone marrow mononuclear cell transplantation for spastic cerebral palsy. J Transl Med. 2017 Feb 24;15(1):48. doi: 10.1186/s12967-017-1149-0. PMID 28235424